CLINICAL TRIAL: NCT00262899
Title: Genetic Counseling for Newly Diagnosed Breast Cancer Patients
Brief Title: Genetic Counseling or Usual Care in Helping Women With Newly Diagnosed Ductal Carcinoma In Situ or Stage I, Stage II, or Stage IIIA Breast Cancer Make Treatment Decisions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marc D Schwartz, Professor of Oncology, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000450155; R01CA108933 (NIH); R01CA074861 (NIH); P30CA051008 (NIH); GUMC-2004-212
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; ductal breast carcinoma in situ; breast cancer in situ; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Counseling; Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid genetic counseling (Experimental): Following randomization, participants will be informed about whether they are assigned to Usual Care (UC) or Rapid Genetic Counseling (RGC). Participants in the UC arm can schedule a genetic counseling appointment at any time during the study if they wish. Participants in the RGC agree to obtain genetic counseling as soon as possible, before they make a definitive surgery decision. RGC can be accomplished by telephone or in-person. The RGC intervention is delivered by highly experienced genetic counselors at each site. This counseling is identical to our standard genetic counseling procedure for newly diagnosed patients. Immediate DNA collection via blood or buccal cell collection is available following counseling. Phone counseling participants will be been mailed a kit for DNA collection or have the option of having the sample collected at at LCCC.
  Interventions: Behavioral: counseling intervention; Other: educational intervention; Procedure: psychosocial assessment and care
- Usual Care (No Intervention): Usual Care (UC) for newly diagnosed breast cancer patients does not typically include a pre-surgical genetic referral. These patients may obtain genetic counseling at their own discretion.

INTERVENTIONS:
Behavioral: counseling intervention
  Arms: Rapid genetic counseling
Other: educational intervention
  Arms: Rapid genetic counseling
Procedure: psychosocial assessment and care
  Arms: Rapid genetic counseling

SUMMARY:
RATIONALE: Genetics education and counseling may help patients make treatment decisions. It is not yet known how genetic counseling or usual care influence patient treatment decisions for breast cancer.

PURPOSE: This randomized clinical trial is studying how well genetic counseling works compared to usual care in helping patients with newly diagnosed ductal carcinoma in situ, stage I, stage II, or stage IIIA breast cancer make treatment decisions.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the impact of rapid genetic counseling (RGC) vs usual care on the medical decisions of women with newly diagnosed ductal carcinoma in situ or stage I-IIIA breast cancer.
* Compare the impact of these interventions on the quality of life and psychological well being of these patients.
* Determine baseline factors that predict who is most and least likely to benefit from RGC in patients undergoing these interventions.
* Compare the cost per quality adjusted life year saved from a societal perspective in patients undergoing these interventions.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating site. Patients are randomized to 1 of 2 interventional arms.

* Arm I (rapid genetic counseling): Patients undergo a 1½ hour genetic counseling session either in person or by telephone. Patients who undergo telephone counseling receive a booklet of visual aids and educational materials. Patient preferences and values are assessed immediately after counseling. Some patients may undergo BRCA1/2 status determination. Patients undergo follow-up telephone interviews at 1, 6, and 12 months.
* Arm II (usual care): Patients receive a packet of breast cancer treatment educational materials. Patient preferences and values are assessed 2 weeks later. Patients undergo follow-up telephone interviews as in arm I.

In both arms, quality of life is assessed at baseline and at 1, 6, and 12 months.

After completion of the study, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 360 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed breast cancer, meeting 1 of the following criteria:

  * Stage 0 disease (ductal carcinoma in situ only)
  * Stage I-IIIA disease
* Must meet 1 of the following criteria:

  * Diagnosis before 50 years of age
  * Diagnosis after 50 years of age AND has 1 of the following:

    * First or second degree relative diagnosed with breast cancer before 50 years of age
    * First or second degree relative diagnosed with ovarian cancer at any age
    * First or second degree relative diagnosed with male breast cancer at any age
* Must not have initiated definitive treatment for breast cancer
* No bilateral, metastatic, or inflammatory breast cancer
* No prior BRCA1/2 counseling or testing
* No prior diagnosis of metastatic cancer of any type
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Surgery

* No prior bilateral mastectomy for breast cancer

Other

* No concurrent treatment for cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2005-08; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Definitive surgery choice as measured by self-reported and medical record verification at 6 months after randomization | 1, 6, and 12 months
Quality of life as measured by functional assessment of cancer therapy for breast cancer (FACT-B) at 1, 6, and 12 months after randomization | 1, 6, and 12 months
Distress as measured by Impact of Events Scale Brief Symptom Inventory at 1, 6, and 12 months after randomization | 1, 6, and 12 months
Knowledge as assessed by Genetic Testing Knowledge Measure at 1 month after randomization | 1 month
Decision outcomes as assessed by Decisional Conflict Scale Satisfaction with Decision Scale at 1 and 6 months after randomization | 1 and 6 months

SECONDARY OUTCOMES:
Cost effectiveness as measured by quality adjusted life years saved at 12 months after randomization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schwartz, PhD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Chevy Chase, Maryland
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Mount Sinai School of Medicine, New York, New York

REFERENCES:
- [Derived] Schwartz MD, Peshkin BN, Isaacs C, Willey S, Valdimarsdottir HB, Nusbaum R, Hooker G, O'Neill S, Jandorf L, Kelly SP, Heinzmann J, Zidell A, Khoury K. Randomized trial of proactive rapid genetic counseling versus usual care for newly diagnosed breast cancer patients. Breast Cancer Res Treat. 2018 Aug;170(3):517-524. doi: 10.1007/s10549-018-4773-3. Epub 2018 Apr 2. PMID 29611029